CLINICAL TRIAL: NCT04835792
Title: Biomarker Study to Evaluate Participants With Previously Treated Lyme Disease in Comparison to Healthy Volunteers
Brief Title: Biomarker Study of Previously Treated Lyme Disease Volunteers in Comparison to Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FlightPath Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FP-LD-001
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Previously Treated for Lyme Disease
  Interventions: Other: Stool and blood collection
- Healthy Volunteers
  Interventions: Other: Stool and blood collection

INTERVENTIONS:
Other: Stool and blood collection — One-time stool and blood collection

SUMMARY:
Non-interventional study evaluating stool and blood samples collected from individuals previously treated with Lyme disease versus healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age.
2. Able to read, understand, and provide signed informed consent.
3. Willing to provide blood and stool samples.
4. Able to communicate adequately and to comply with the requirements for the entire study.
5. Must be willing to discontinue antibiotics 2 weeks prior to sample collection.
6. If participating in the previously treated Lyme Disease arm, the participants must meet the following criteria: 1) Diagnosis of prior Lyme Disease supported by either an erythema migrans rash (either classic "bull's eye" or irregular) OR a CDC-positive Western blot, 2) previously treated with antibiotics for Lyme Disease, 3) remains ill six months or more after receiving preliminary treatment with antibiotics for Lyme disease (e.g., fatigue, musculoskeletal pain, or neurocognitive symptoms).
7. If participating in the healthy volunteer arm, the participants must meet the following criteria: 1) must not have had a Lyme Disease diagnosis, 2) in generally good health

Exclusion Criteria:

1. Unwilling or unable to comply with the protocol (e.g., scheduled visits, laboratory tests, other study procedures, and study restrictions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Previously treated Lyme disease volunteers and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
• To evaluate and compare the microbiome of normal participants and participants with previously treated Lyme Disease | 30 days
• To evaluate and compare the transcriptome of normal participants and participants with previously treated Lyme Disease | 30 days
• To evaluate and compare the metabolome of normal participants and participants with previously treated Lyme Disease | 30 days
• Evaluation of symptoms and prior medications/treatments of normal participants and participants with previously treated Lyme Disease | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Curtis Scribner, Berkeley, California, United States